CLINICAL TRIAL: NCT01250782
Title: Effectiveness of Dipeptide N (2)-L-Alanyl-L-Glutamine in Trauma ICU Patients: Pilot, Prospective, Randomized and Double Blind Study.
Acronym: GluTrac
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Son Dureta (Other)
Responsible Party: Pedro Marsé-Milla, Hospital Universitari Son Dureta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GlnHSD-001-09
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Trauma ICU Patients
Keywords: Glutamine, trauma patients, infections, mortality
MeSH Terms: conditions — Infections | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiological Serum (Placebo Comparator)
  Interventions: Drug: Physiological serum
- Glutamine (Active Comparator)
  Interventions: Drug: Glutamine

INTERVENTIONS:
Drug: Glutamine — 0.5 g/kg/day of dipeptide N (2)-L-Alanyl-L-Glutamine
  Arms: Glutamine
Drug: Physiological serum — 100 mL of physiological serum indistinguishable from active comparator
  Arms: Physiological Serum

SUMMARY:
Recent reports suggest that most beneficial results of glutamine have been obtained with the parenteral administration of high doses of glutamine (0.35 g/Kg/d) and in some special group of patients, such as traumatic patients. Nevertheless total parenteral nutrition is not often used in critically ill patients.

The endovenous administration of the the dipeptide N(2)-L-alanyl-L-glutamine in trauma ICU patients can reduce the number of infections, ICU length of stay and mortality.

This benefit can be achieved independently the type of nutrition (enteral or parenteral nutrition), being a pharmaconutrient.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of the endovenous administration endovenous glutamine to reduce the number of infectious complications, mortality and ICU length of stay in trauma ICU patients. To achieve this objective we have designed this pilot study to obtain the necessary data to design a bigger trial in the future.

Other objectives include:

* To evaluate the efficacy of glutamine in different patients regarding their severity: patients with an Injury Severity Score> 25 and patients with lower plasma levels of glutamine.
* To registry the possible adverse events of the endovenous administration of glutamine.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe trauma, as defined by an Injury Severity Score (ISS) > 10 points were included in the study.
* Traumatic patients who required enteral or parenteral nutrition during the first 48 hours after hospital admission
* Written informed consent

Exclusion Criteria:

* patients whose life expectancy was less than 5 days,
* who were allergic to glutamine,
* Patients included in any other trial
* Cirrhotic patients (Child C)
* Chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Number of infections | ICU discharge (median ten days)
  Based on the results of the ENVIN trial, the median ICU length of stay of trauma patients admitted to the ICU in Spain, is 10 days.

SECONDARY OUTCOMES:
ICU Mortality | ICU mortality measured at 1 month after hospital admission
SAfety of endovenous administration | 5 days from the beginning of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Son Dureta, Palma, Balearic Islands, Spain